CLINICAL TRIAL: NCT04809480
Title: The Impact of COVID-19 Outbreak on The Incidence of Acute Invasive Fungal Rhinosinusitis
Brief Title: COVID-19 and Acute Invasive Fungal Rhinosinusitis
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdulkarim Hasan, laboratory manager, Al-Azhar University
Other Study IDs: 20- 11- 002
Record Dates: First submitted 2021-03-19; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: fungal sinusitis; rhinosinusitis
MeSH Terms: conditions — COVID-19; Rhinosinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-COVID19 patients: All acute invasive fungal rhinosinusitis patients managed in our hospital from January 2017 up to February 2020
  Interventions: Diagnostic Test: Fungal rhinosinusitis
- COVID19 patients: All acute invasive fungal rhinosinusitis patients managed in our hospital from February 2020 up to December 2020 with positive COVID19 PCR test
  Interventions: Diagnostic Test: Fungal rhinosinusitis

INTERVENTIONS:
Diagnostic Test: Fungal rhinosinusitis — Pathology examination

SUMMARY:
Data for acute invasive rhinosinusitis was obtained from the Otorhinolaryngology departments at our tertiary hospital at the period from January 2017 to December 2020. Then the risk factors of comorbid diseases and fungal types between post-Covid-19 and non-Covid-19 groups regarding the incidence of invasive rhinosinusitis are compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age and sex. invasive rhinosinusoitis diagnosis based on clinical , endoscopic diagnosis
* Positive findings for acute sinusitis on sinus computed tomography (CT) scan in addition to fungal determination by histopathological examination of specimen of affected tissues for detection of the type of fungi.
* Positive PCR was confirmed from the patient's files at the isolation hospitals for COVID 19 group.

Exclusion Criteria:

* Patients who completed management outside our hospital

Ages: 15 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any age and sex medically managed in AlAzhar Hospitals in Egypt for invasive rhinosinusoitis
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Fungus detection | 2 weeks
  Culture and microscopic examination by the light microscope to examine the different types of the fungi using hematoxylin & eosin stain and Periodic acid-Schiff stain which is positive in fungi

IPD SHARING:
Plan to Share IPD: Undecided
publication in medical journal